CLINICAL TRIAL: NCT01935362
Title: Bioavailability of Flavanones Compounds and Their Impact on Cardiovascular Health
Brief Title: Impact of Oranges on Cardiovascular Health
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Dr Andrea Day and Prof Gary Williamson (Unknown)
Responsible Party: Principal Investigator, Abdurrahman M Sweidan, Mr, University of Leeds
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: MEEC 12-025
Record Dates: First submitted 2013-08-20; First posted 2013-09-05 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Blood Pressure; Endothelial Dysfunction; Cardiovascular Disease Risk Reduction
Keywords: Flavanones; Bioavailability; Blood vessel health; Blood glucose

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): Placebo administered to participant
  Interventions: Dietary Supplement: Placebo
- Citrus supplement (Active Comparator): Citrus supplement administered to participant
  Interventions: Dietary Supplement: Citrus supplement

INTERVENTIONS:
Dietary Supplement: Citrus supplement
  Arms: Citrus supplement
Dietary Supplement: Placebo
  Arms: placebo

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of deaths in the Western world. Established risk factors include high LDL cholesterol, high blood pressure and diabetes. Poor blood vessel health is considered a predictor of future CVD risk, but can be reversed. Several different measurements can be used to determine blood vessel health; such as blood pressure (BP), and newer techniques which measure blood flow through the arteries after a blood pressure cuff restricts blood flow for a few minutes in one arm.

Flavonoids are compounds found in plant-based foods, and are associated with a reduced risk of CVD. From the previous studies, there is strong evidence that orange juice and citrus foods which have higher amount of specific citrus flavonoids improved cardiovascular risk factors such as BP and blood vessel health. Absorption of citrus flavonoids occurs in the colon after bacteria breakdown the forms found in food. After the flavonoids are absorbed into the blood they are modification by liver enzymes before they are excreted in the urine. A large range of citrus flavonoid have been found excreted in the urinary, ranging anywhere from 0-57% of the dose. Variation in the potential health effect may reflect the level of the citrus flavonoid absorbed, and this is not often considered in human studies.

This study is a 4-week double-blinded, randomized, cross-over intervention trial using a commercially-available orange juice supplement and a placebo control. The aims of the study are to determine whether orange juice supplements reduce blood pressure and improve blood vessel health after 4 weeks. Furthermore, to determine if there is a relationship between absorption of flavonoids (as measured by urinary excretion) and changes in blood pressure or blood vessel health.

The participants will need to attend 4 sessions on 4 separate study days, every 4 weeks for 12 weeks. On each study day they will have their weight, height, waist circumference, and blood pressure measured. A finger-prick blood sample, using a single-use lancet (Accu-Chek Safe T Pro Plus), will be taken to check the fasting blood glucose level. Blood flow in fingertips will be monitored before and after reducing blood flow in your forearm using a blood pressure cuff (called an EndoPAT). Participants will be asked to collect urine for 24 hr on each of the study days, and to consume the supplements provided daily for two sets of 4 weeks (there will be 4 weeks in the middle without any supplements).

An improvement in blood pressure and/or blood flow will provide evidence that blood vessel health has improved through short-term (4 week) use of a citrus flavonoid supplement

ELIGIBILITY:
Inclusion Criteria:

* No known cardiovascular disease or diabetes
* Age between 30-60 years
* Heavier than average (Body mass index, BMI ≥ 25 kg/m2)
* Currently non smoker
* Willing to consume orange juice supplements for 2 months
* Male and female are equally eligible as not mentioned on advert

Exclusion Criteria:

* Those who Taken any antibiotics in the 2 months prior to the study
* Those who consume dietary or herbal supplements
* previous surgery on gastrointestinal tract
* Those who currently taking medication
* Current smokers, or ex-smokers ceasing < 3 months ago
* pregnant or breast feeding
* Those with known allergies to the intervention treatment

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-06; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
blood pressure | Baseline and 4 weeks
  Change in systolic and diastolic blood pressure
An improvement in blood flow | Baseline and 4 weeks
  Change in blood flow using Endo-PAT device

SECONDARY OUTCOMES:
blood glucose | Baseline and 4 weeks
  Change in blood glucose level in plasma,
bioavailability of flavanones compounds | Baseline and 4 weeks
  Change of urine flavanones from the baseline and after 4 weeks of each arm

CONTACTS AND LOCATIONS:
Overall Officials: Abdurrahman M Sweidan, Principal Investigator — University of Leeds
Locations (1):
- School Of Food Science and Nutrition, University Of Leeds, Leeds, West Yorkshire, United Kingdom

REFERENCES:
- See also: Click here for more information about this study: Impact of oranges on cardiovascular health — http://www.food.leeds.ac.uk/orangejuice